CLINICAL TRIAL: NCT01043510
Title: A Trial Investigating the Pharmacodynamic and Pharmacokinetic Properties of NN1250 at Steady State Conditions in Subjects With Type 2 Diabetes of Different Race and/or Ethnicity
Brief Title: The Effect of NN1250 in Subjects With Type 2 Diabetes of Different Race and/or Ethnic Origin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1250-3762; U1111-1112-6185 (Other: WHO)
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec; Insulin Detemir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A1, first period (Experimental)
  Interventions: Drug: insulin degludec
- A2, second period (Active Comparator)
  Interventions: Drug: insulin detemir
- B1, first period (Active Comparator)
  Interventions: Drug: insulin detemir
- B2, second period (Experimental)
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec — 0.6 U/kg body weight injected subcutaneously (under the skin), once daily for 6 days
  Arms: A1, first period; B2, second period
Drug: insulin detemir — 0.6 U/kg body weight injected subcutaneously (under the skin), once daily for 6 days
  Arms: A2, second period; B1, first period

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to investigate the pharmacodynamic (effect) and pharmacokinetic (exposure of drug) properties of NN1250 (insulin degludec, IDeg) in subjects with type 2 diabetes of different race and/or ethnicity.

ELIGIBILITY:
Inclusion Criteria:

* Either - Black or African American not of Hispanic or Latino origin or - White of Hispanic or Latino origin or - White not of Hispanic or Latino origin
* Type 2 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Treated with insulin for at least 3 months, alone or in combination with maximum 2 oral antidiabetic drugs (OADs)
* Body mass index maximum 40.0 kg/m^2

Exclusion Criteria:

* Use of GLP-1 receptor agonists (exenatide, liraglutide), thiazolidinediones or dipeptidyl peptidase-4 (DPP-4) inhibitors within 3 months prior to screening
* History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction
* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate curve during one dosing interval at steady state | 0-24 hours (derived on treatment day 6)

SECONDARY OUTCOMES:
Area under the Insulin Degludec concentration-time curve during one dosing interval at steady state | 0-24 hours (derived on treatment day 6)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Chula Vista, California, United States

REFERENCES:
- [Result] Hompesch M, Morrow L, Watkins E, Roepstorff C, Thomsen HF, Haahr H. Pharmacokinetic and pharmacodynamic responses of insulin degludec in African American, white, and Hispanic/Latino patients with type 2 diabetes mellitus. Clin Ther. 2014 Apr 1;36(4):507-15. doi: 10.1016/j.clinthera.2013.12.014. Epub 2014 Feb 5. PMID 24508419
- [Result] Heise T, Korsatko S, Nosek L, Coester HV, Deller S, Roepstorff C, Segel S, Kapur R, Haahr H, Hompesch M. Steady state is reached within 2-3 days of once-daily administration of degludec, a basal insulin with an ultralong duration of action. J Diabetes. 2016 Jan;8(1):132-8. doi: 10.1111/1753-0407.12266. Epub 2015 Mar 24. PMID 25581159
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com